CLINICAL TRIAL: NCT03519503
Title: Promoting Infant Health and Nutrition in Sub-Saharan Africa (PROMISE): Safety and Efficacy of Infant Peri-Exposure Prophylaxis (PEP) to Prevent HIV-1 Transmission by Breastfeeding Mechanisms & Safety (M&S)
Brief Title: Infant Peri-Exposure Prophylaxis to Prevent HIV-1 Transmission by Breastfeeding: Mechanisms & Safety
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS 12341 PROMISE-PEP M&S
Record Dates: First submitted 2017-11-02; First posted 2018-05-09 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Growth and Development
Keywords: HIV; Neuropsychological tests; PMTCT; PreP

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
General objective

* To assess the long-term safety and efficacy of one-year infant prophylaxis using lamivudine (3TC) or lopinavir/ritonavir (LPV/r) to prevent post-natal transmission through breastfeeding.
* To investigate the biological mechanisms involved in postnatal HIV transmission.

Specific objectives

* To compare the long-term safety of infant prophylaxis using either 3TC versus LPV/r on child development (growth, somatic and mental health), mortality, adrenal function, liver function, full blood count and mitochondrial toxicity.
* To estimate the final efficacy data of 50 weeks of infant prophylaxis using either LPV/r or 3TC, since some mothers may have resumed breastfeeding after the trial.
* To profile miRNA in breast milk according to maternal HIV status and HIV transmission.
* To determine the influence of maternal milk on infant gut inflammation in an in vitro 3D-intestinal model (CACO-2 cells).

The study population will comprise all ANRS 12174 PROMISE-PEP trial participants who completed the 50 week follow-up and are not HIV infected. An estimate of 881 mother-child pairs from the ANRS 12174 PROMISE- PEP will be recruited.

This study is structured in two parts. The 'clinical & biological safety' component involves a cross sectional survey. A clinical and neuropsychological examination of participants will be conducted. In addition one venous blood sample will be collected to evaluate children HIV status, full blood count, liver & adrenal function and mitochondrial toxicity. Capillary hair follicles will be collected from 100 children in Zambia to study their genome integrity.

The 'mechanisms' component includes biological assays to be conducted on breast milk samples previously collected from HIV infected, transmitting or non-infected mothers enrolled at ANRS 12174 PROMISE-PEP trial.

Primary endpoint: Long term survival, mortality rate, measurements of infant growth (length and weight), somatic and neuropsychological development of the 5 year old children enrolled in the ANRS 12174 PROMISE- PEP trial.

Secondary endpoints: HIV seroconversion since last PROMISE PEP trial visit, full blood count, liver function, adrenal function, serum lactate. Number of mitochondrial DNA copies per cell & percentage of mitochondrial DNA deletion for mitochondrial toxicity. Number of micronuclei & number of Ɣ-tubulin spot per cell to study genomic toxicity.

DETAILED DESCRIPTION:
Background Besides optimal efficacy, Prevention of mother-to-child transmission of HIV(PMTCT) strategies must have a very good safety profile (1). Indeed, very large quantities of children will be exposed to these strategies, and the vast majority of them will not eventually be infected. Because in utero HIV exposure followed by one year of antiretroviral treatment (i.e at the time of infant embryogenesis and maturation) may have long-term consequences, such as hampering child development, an evaluation of safety beyond the end of prophylaxis is necessary to get a comprehensive knowledge of the true benefits/risks balance of PMTCT strategies.

A recent review of the state of the art identified several knowledge gaps in the current understanding of Mother To Child Transmission (2). The role of HIV breast milk cell reservoirs in the HIV transmission through breastfeeding is still unclear. The effect of immune factors present in breast milk of HIV infected mothers on HIV population dynamics is also unknown as well as the permeability of infant's gut mucosa and the mechanisms involved on HIV transmission.

The ANRS 12174 randomized controlled trial (ClinicalTrials.gov Identifier: NCT00640263) evaluated 3TC and LPV/r as infant Prep drugs for 50 weeks in HIV uninfected babies at day 7, with monthly follow-up. In addition, breast milk samples were collected four times during follow-up with infant plasma and cell pellets collected at weeks 6, 22 and 38, and infants Dried Blood Spots (DBS) every 3 months. The final results showed that both 3TC and LPV/r achieved very low rates of transmission with an excellent clinical tolerance and no difference between arms in terms of efficacy or safety. In total, 1103 infants completed the final visit.

This study presents a unique opportunity to i) investigate the mechanisms of HIV-1 post-natal transmission, iii) to assess long-term safety of LPV/r and 3TC and ii) to estimate the final efficacy of infant peri-exposure prophylaxis (PreP), since some children were still exposed at the end of the study.

The study will be conducted at the four ANRS 12174 PROMISE-PEP trial sites, namely East London (South Africa), Ouagadougou (Burkina Faso), Lusaka (Zambia) and Mbale (Uganda).

Clinical and Biological safety component At enrolment, children will be assessed for hospitalisation events since the end of the ANRS 12174 PROMISE-PEP trial, mortality rate, growth, neurodevelopment, mitochondrial and genomic toxicity, and blood biochemical parameters such as full blood count, liver function and the level of adrenal hormones. All biological assays and explorations in this study will be carried out blindly, Mitochondrial DNA depletion study: DBS will be collected from all children at enrolment. Samples will be randomized and only 50 samples from Burkina Faso, Uganda and Zambia will be analysed (N=150) as it give us enough power to detect the statistical inferences within the population.

Genome integrity study:The genome integrity assessment will include 50 children from each of the two PROMISE-PEP arms selected by randomization. (n=100 in total). The Zambian site is the only one with the necessary expertise and laboratory equipment for freezing cells. Therefore, the genome integrity study will only be conducted at this site. As a source of adherent cells, plucked hairs will be collected and frozen in 10% dimethylsulfoxide (DMSO) solution.

Children will be assessed through a battery of tests; the Kaufman Assessment Battery for Children - Second edition (KABC-II), the Movement Assessment Battery for Children - Second Edition (M-ABC2), the Test of Variables of Attention (TOVA)-visual, the Strengths and Difficulties Questionnaire (SDQ25) designed to evaluate the main neuropsychological domains considered to be affected in HIV pediatric disease. Children will be evaluated when they are over 5 years of age.

The 'mechanisms' component includes biological assays to be conducted on breast milk samples previously collected from HIV infected, transmitting or not transmitting mothers enrolled at ANRS 12174 PROMISE-PEP trial. Two studies will be conducted.

* The first study will investigate the specific microRNAs found in exosomes present in breast milk that are linked to regulation immune pathways. We propose to investigate the different miRNA profile in human breast milk in correlation to HIV status and HIV transmission. We also hypothesize that the involved pathways on may be linked with the local mucosal immunity of the mother breast but also with the gut mucosal immunity of the recipient child.
* The second study will focus on the effect of breast milk effect on the cytokine profile of infant's intestinal cells. We aim to determine 1/ the enterocyte cytokine profile exposed to breast milk compounds; 2/ the influence of milk on the transcytosis of T-lymphocytes, both HIV-infected and HIV negative.

ELIGIBILITY:
Inclusion Criteria:

* Having taken part in the ANRS 12174 PROMISE-PEP trial until the final (50 week) visit;
* Not being infected with HIV during the duration of the ANRS 12174 PROMISE-PEP trial.

Exclusion Criteria:

* Parent refusal to participate in the study after information about the PROMISE M&S project is given.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will comprise all ANRS 12174 PROMISE-PEP trial participants who completed the 50 week follow-up and are not HIV infected. There are 1101 children fulfilling the inclusion criteria over the four African sites with an estimation of 80% of them being recruited on PROMISE M&S study (N=881).
Sampling Method: Non-Probability Sample
Enrollment: 562 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
HIV seroconversion | From date of last visit in PROMISE PEP study (week 50 of follow-up) until the date of PROMISE-PEP M&S inclusion visit, assessed up to 96 months
  Number of children with positive HIV test

SECONDARY OUTCOMES:
Long term survival | From date of last visit in PROMISE PEP study (week 50 of follow-up) until the date of first documented date of death from any cause, assessed up to 96 months
  Time to death
Mortality rate | From date of last visit in PROMISE PEP study (week 50 of follow-up) until the date of first documented date of death from any cause, assessed up to 96 months
  Number of deaths
Height | Cross-sectional survey during the inclusion visit
  measured in centimeters
Weight | Cross-sectional survey during the inclusion visit
  measured in kilograms
Infant growth | Cross-sectional survey during the inclusion visit
  weight-for-height, height for age, weight for age and body mass index for age measured by Z-scores
Neuro-psychological development | Cross-sectional survey during the inclusion visit
  Development measured by M-ABC2, KABC-II, SDQ25 and TOVA-visual total standard test scores, percentiles, age specific norms and standard deviations.
Biological disorders | Cross-sectional survey during the inclusion visit
  Number of children with normal full blood count
Biological disorders | Cross-sectional survey during the inclusion visit
  Number of children with normal liver function tests
Biological disorders | Cross-sectional survey during the inclusion visit
  Number of children with normal functioning of adrenal glands
Biological disorders | Cross-sectional survey during the inclusion visit
  Number of children with normal serum lactate levels

OTHER OUTCOMES:
Mitochondrial toxicity | Cross-sectional survey during the inclusion visit
  Number of mitochondrial DNA copies per cell
Mitochondrial toxicity | Cross-sectional survey during the inclusion visit
  Percentage of mitochondrial DNA deletion
Genome integrity | Cross-sectional survey during the inclusion visit
  Number of micronuclei
Genome integrity | Cross-sectional survey during the inclusion visit
  Number of Ɣ-tubulin spot per cell

CONTACTS AND LOCATIONS:
Overall Officials: Chipepo KANKASA, MD, PhD, Principal Investigator — University of Zambia; Mandisa SINGATA, PhD, Principal Investigator — University of Fort Hare, South Africa; Nicolas MEDA, MD, PhD, Principal Investigator — University of Ouagadougou, Burkina Faso; James K TUMWINE, MD,PhD, Principal Investigator — University of Makerere, Uganda
Locations (4):
- Centre Hospitalier Universitaire Blaise Compraore, Ouagadougou, Burkina Faso
- Cecilia Makiwane hospital, East London, South Africa
- PROMISE M&S site, Mbale, Uganda
- Paediatric Center Of Excellence, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heidari S, Mofenson L, Cotton MF, Marlink R, Cahn P, Katabira E. Antiretroviral drugs for preventing mother-to-child transmission of HIV: a review of potential effects on HIV-exposed but uninfected children. J Acquir Immune Defic Syndr. 2011 Aug 1;57(4):290-6. doi: 10.1097/QAI.0b013e318221c56a. PMID 21602695
- [Background] Van de Perre P, Rubbo PA, Viljoen J, Nagot N, Tylleskar T, Lepage P, Vendrell JP, Tuaillon E. HIV-1 reservoirs in breast milk and challenges to elimination of breast-feeding transmission of HIV-1. Sci Transl Med. 2012 Jul 18;4(143):143sr3. doi: 10.1126/scitranslmed.3003327. PMID 22814853
- [Background] Nagot N, Kankasa C, Tumwine JK, Meda N, Hofmeyr GJ, Vallo R, Mwiya M, Kwagala M, Traore H, Sunday A, Singata M, Siuluta C, Some E, Rutagwera D, Neboua D, Ndeezi G, Jackson D, Marechal V, Neveu D, Engebretsen IMS, Lombard C, Blanche S, Sommerfelt H, Rekacewicz C, Tylleskar T, Van de Perre P; ANRS 12174 Trial Group. Extended pre-exposure prophylaxis with lopinavir-ritonavir versus lamivudine to prevent HIV-1 transmission through breastfeeding up to 50 weeks in infants in Africa (ANRS 12174): a randomised controlled trial. Lancet. 2016 Feb 6;387(10018):566-573. doi: 10.1016/S0140-6736(15)00984-8. Epub 2015 Nov 19. PMID 26603917